CLINICAL TRIAL: NCT03251989
Title: Exploring Outcomes and Risk in Patients With Rare Central Nervous System Tumors
Brief Title: Rare CNS Tumors Outcomes &Risk
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917141; 17-C-N141
Record Dates: First submitted 2017-08-15; First posted 2017-08-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12-02

CONDITIONS: High Grade Meningioma; Ependymoma; Medulloblastoma; PNET; Primary CNS Sarcoma
Keywords: Brain Tumor; Central Nervous System Tumors; Choroid Plexus Tumors; Gliomas; Atypical Teratoid Rhabdoid Tumor; Natural History
MeSH Terms: conditions — Ependymoma; Medulloblastoma; Neuroectodermal Tumors, Primitive; Brain Neoplasms; Central Nervous System Neoplasms; Choroid Plexus Neoplasms; Glioma; Rhabdoid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Patient with a rare CNS diagnosis: A diagnosis of rare CNS Tumors

SUMMARY:
Background:

Primary tumors of the brain and spine are those that start in the brain or spine. These tumors are rare, accounting for <2% of all cancers diagnosed in the United States. Some of these tumors occur in less than 2,000 people per year. Researchers want to study a large group of people with this kind of tumor. They want to learn more about the tumors, including the risk factors related to how they develop in adults.

Objective: To collect health and gene data to learn about what changes are associated with a rare CNS Tumors, to eventually screen for these changes or target the genes in treatment.

Eligibility: Adult participants >= 18 years of age who self- identify as being diagnosed with one of 12 rare CNS tumors, including: Atypical teratoid rhabdoid tumor (ATRT); Brainstem and midline gliomas; Choroid plexus tumors; Ependymoma; High grade meningioma; Gliomatosis cerebri; Medulloblastoma; Oligodendroglioma / Anaplastic oligodendroglioma; Pineal region tumors; Pleomorphic xanthroastrocytoma / Anaplastic pleomorphic xanthroastrocytoma; PNET (Supratentorial embryonal tumor); Primary CNS sarcoma / Secondary CNS sarcoma (Gliosarcoma).

Design:

Participants will be invited to participate through an ad on the CERN Foundation website (ependymoma), information on the Neuro-Oncology Branch website and other identified advocacy and social media sites and direct mailer to those who have already participated in the EO projects. (Registered Trademark)

* Interested participants will complete an enrollment form that will be sent to the study coordinator.
* The coordinator will then send the participant a consent form and schedule a time for phone consent.
* Participants will complete the Rare CNS tumors Outcomes Survey and once completed, the Rare CNS tumors Risk survey. (Registered Trademark)
* The questions on the Outcomes Survey will include treatment history, symptoms social and clinical information and it should take about 25-35 minutes. The Risk survey will cover their demographic information, personal medical history, family medical history and environmental exposures. This should take about 52 minutes.
* Participants who have physical problems can have help with the surveys and forms.
* Once the surveys are completed, participants will be mailed a kit to collect saliva for germline DNA. Participants will ship the sample to the study team in a prepaid envelope
* If the sample is not sufficient, participants will be contacted to give provide an additional sample.

DETAILED DESCRIPTION:
Background:

Rare cancers are defined as those with <40,000 cases per year. There are over 130 separate types of primary CNS tumors, all of which meet the definition of a rare cancer. However, some CNS cancers have incidences of less than 1,000 cases per year. Because of its relative rarity, limited reports of the presentation and clinical course have been completed. With the support of the CERN-Foundation, the Adult Ependymoma Outcomes Projects (AEO) was launched to address this lack of information for one type of rare CNS tumor- ependymoma. Using an online platform, participants and families from across the world have participated, providing information that has helped elucidate the presentation and ongoing health of individuals with this disease. To date, over 300 adults have participated with over 95% reporting interest in continuing and expanding their participation. Results from the AEO baseline survey and a follow-up survey (AEOII addressing socioeconomic impact of the disease) have been published. The most recent data from the AEO has been presented at the Society for Neuro-Oncology (SNO) annual meetings in 2015 and 2016.

An additional consequence of the relative rarity of these CNS tumors, studies to evaluate risk factors for the occurrence of these rare CNS tumors or predicting the clinical course of these rare CNS tumors are also limited. Rare CNS tumors like other cancers, occur when there are changes to genes that control the way cells grow and divide often as a result of exposure to other environmental risk factors. Therefore, exploring genetic changes in persons with rare CNS tumors will allow us to begin to understand what changes are associated specifically with these tumors. To date, these participants are often included as part of larger cohorts which include other types of brain tumors. We now understand that even among gliomas, the risk factors differ. Therefore, identifying the risk factors specifically associated with rare CNS tumors is critical for primary prevention and early detection. This knowledge would allow scientists and physicians to eventually screen for these changes or target the genes or the processes they control for treatment purposes.

Objectives:

The primary objectives of this study are to:

* Obtain self-reported data on treatment, symptoms, functional status, and quality of life for adult participants with rare CNS tumors.
* To evaluate the relationship between health status and disease and treatment characteristics.
* To evaluate self-reported clinical and demographic risk factors in adult participants in the rare CNS tumor participant population.
* To explore genomic susceptibility in participants with rare CNS tumors

Eligibility:

The adult rare CNS tumor population for this study are participants >= 18 years of age who self- identify as being diagnosed with one of 12 rare CNS tumors, including:

* Atypical teratoid rhabdoid tumor (ATRT)
* Brainstem and midline gliomas
* Choroid plexus tumors

  * Choroid plexus carcinoma
  * Choroid plexus papilloma
  * Atypical choroid plexus papilloma
* Ependymoma

  * Subependymoma
  * Myxopapillary ependymoma
  * Papillary ependymoma
  * Clear cell ependymoma
  * Tanycytic ependymoma
  * RELA fusion-positive
  * Anaplastic ependymoma
  * Posterior Fossa A
  * Posterior Fossa B
* High grade meningioma

  * Chordoid meningioma
  * Clear cell meningioma
  * Atypical meningioma
  * Papillary meningioma
  * Rhabdoid meningioma
  * Anaplastic (malignant) meningioma
* Gliomatosis cerebri
* Medulloblastoma

  * Sonic Hedge Hog (SHH)
  * WNT
  * Group 3
  * Group 4
* Oligodendroglioma / Anaplastic oligodendroglioma
* Pineal region Tumors

  * Pineoblastoma
  * Pineocytoma
  * Pineal parenchymal tumor of intermediate differentiation
  * Papillary tumor of the pineal region
* Pleomorphic xanthroastrocytoma / Anaplastic pleomorphic xanthroastrocytoma
* PNET (Supratentorial embryonal tumor)
* Primary CNS sarcoma / Secondary CNS sarcoma (Gliosarcoma)

Design:

* This study represents an ongoing effort to systematically evaluate outcomes in a large group of participants with these rare tumors. It will provide descriptive data which can be used to design further studies evaluating interventions related to identified health and quality of life related issues for this participant population.
* Participants will be invited to participate through an ad on the CERN Foundation website (ependymoma), information on the Neuro-Oncology Branch website and other identified advocacy and social media sites and direct mailer to those who have already participated in the EO projects.
* The goal of adding the Rare CNS tumors Risk Survey is to implement a survey to further evaluate participants in the EO for several known and suspected risk factors for rare CNS tumors and to obtain germline DNA to interrogate genomic susceptibility to the disease.
* Interested participants will complete an enrollment form that will be sent to the study coordinator. Once submitted, the study coordinator will then send the participant a consent form and schedule a time for remote consent if interested.
* Once consent is obtained, the study coordinator will send the participant instructions and a unique link that they will use to access and complete the survey(s).
* Once the surveys are completed, the study coordinator will email the participant a request for medical records to help us collect more health information related to the care of their Rare CNS tumor diagnosis.
* Once the survey(s) are completed, the participant will be mailed a kit to collect saliva for germline DNA.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants with rare CNS tumors who meet the following criteria will be invited to participate in the study:

* A diagnosis of rare CNS tumors, (Atypical teratoid rhabdoid tumor (ATRT); Brainstem and midline gliomas; Choroid plexus tumors; Ependymoma; High grade meningioma; Gliomatosis cerebri; Medulloblastoma; Oligodendroglioma / Anaplastic oligodendroglioma; Pineal region tumors; Pleomorphic xanthroastrocytoma / Anaplastic pleomorphic xanthroastrocytoma; PNET (Supratentorial embryonal tumor); Primary CNS sarcoma / Secondary CNS sarcoma (Gliosarcoma) or as reported by the participant:
* Participants who are currently >= 18 years of age with the initial rare CNS tumor diagnosis occurring at any point in their lifetime are eligible.
* Ability to speak, write, and read English, as questionnaires available in English language only.
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA: See inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be solicited through the Collaborative Ependymoma Research Network (CERN), information on the Neuro-Oncology Branch website and other advocacy organization websites, mailing list and social media sites.@@@
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Relationship between health status and disease and treatment characteristics as well as clinical and demographic risk factors as self reported by adult participants with rare CNS tumors; and the relationship of genomic susceptibility of the popu... | completion of study
  Obtain self-reported data on treatment, symptoms, functional status, and quality of life for adult participants with rare CNS tumors To evaluate the relationship between health status and disease and treatment characteristics. To evaluate self-reported clinical and demographic risk factors in adult participants in the rare CNS tumors participant population. To explore genomic susceptibility in participants with rare CNS tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Tito R Mendoza, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI)/ Neuro-Oncology Branch, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active. @@@@@@All collected IPD will be available after primary analysis have been published.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Armstrong TS, Vera-Bolanos E, Gilbert MR. Clinical course of adult patients with ependymoma: results of the Adult Ependymoma Outcomes Project. Cancer. 2011 Nov 15;117(22):5133-41. doi: 10.1002/cncr.26181. Epub 2011 Apr 28. PMID 21538344
- [Background] Walbert T, Mendoza TR, Vera-Bolanos E, Acquaye A, Gilbert MR, Armstrong TS. Symptoms and socio-economic impact of ependymoma on adult patients: results of the Adult Ependymoma Outcomes Project 2. J Neurooncol. 2015 Jan;121(2):341-8. doi: 10.1007/s11060-014-1638-4. Epub 2014 Oct 31. PMID 25359395
- [Background] Acquaye AA, Vera E, Gilbert MR, Armstrong TS. Clinical presentation and outcomes for adult ependymoma patients. Cancer. 2017 Feb 1;123(3):494-501. doi: 10.1002/cncr.30355. Epub 2016 Sep 28. PMID 27679985
- [Derived] McIver BA, Davis TS, Reinhart K, Vera E, Acquaye-Mallory A, Choi A, Kunst T, Johnson M, Grajkowska E, Miller H, Reyes J, Gilbert MR, Armstrong TS, Wright ML. Evaluating Clinical and Sociodemographic Risk for Symptom Burden Associated Interference With Daily Functioning in the Primary Brain Tumor Patient Population. Cancer Med. 2025 Mar;14(5):e70682. doi: 10.1002/cam4.70682. PMID 40052556